CLINICAL TRIAL: NCT01529203
Title: Subjects' Satisfaction on Pan Facial Aesthetic Enhancement After Treatment With Azzalure® and the Restylane® Range
Acronym: FIRST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RD.03.SPR.29097
Record Dates: First submitted 2012-01-30; First posted 2012-02-08 (Estimated); Results first posted 2014-04-25 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2014-09

CONDITIONS: Aging
MeSH Terms: interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azzalure and Restylane (Other): All subjects will be injected with Azzalure and Restylane
  Interventions: Drug: Botulinum Toxin Type A (Azzalure); Device: Restylane ranges

INTERVENTIONS:
Drug: Botulinum Toxin Type A (Azzalure) — Powder for solution for injection
Device: Restylane ranges — Hyaluronic acid (HA) 20 mg/mL + Lidocaine 0.3% (Restylane® Lidocaine, Restylane® Perlane™ Lidocaine, Restylane® SubQ Lidocaine, Restylane® Lip Volume, Restylane® Lip Refresh)

SUMMARY:
The aim of this study is to assess subjects' satisfaction linked to the pan facial management of rejuvenation with injections of Azzalure® and Restylane® fillers.

This will be an open, multi-centre study.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female subjects, aged 18 to 64 years, seeking treatment for correction of dynamic wrinkles of the upper third of the face and correction of facial volume loss, and meeting other specific eligibility criteria

Main Exclusion Criteria:

* Female subject who is pregnant, nursing or planning a pregnancy during the study
* Subject with any contraindications to the injection of hyaluronic acid (see package inserts)
* Subject with any contraindications to the injection of botulinum toxin (see package insert)
* Subject with a personal history of allergic/anaphylactic reactions including hypersensitivity to crossed-linked hyaluronic acid or botulinum toxin
* Concurrent treatment that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of at least one of the study treatments
* Subject with a history of dissatisfaction with facial aesthetic procedures involving dermal implant injections or subject with unattainable expectations
* Subject currently enrolled in another investigational study or who participated in such a study in the past 30 days prior to baseline visit

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- France (2):
  - Galderma investigational site, Bordeaux
  - Galderma investigational site, Metz
- Galderma investigational site, Madrid, Spain
- United Kingdom (2):
  - Galderma investigational site, London
  - Galderma investigational site, Street

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Azzalure and Restylane
Started | 60
Completed | 57
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Azzalure and Restylane
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (7.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 60
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  France | 20
  Spain | 20
  United Kingdom | 20

OUTCOME MEASURES:

1. Primary Outcome: Subject Satisfaction for the Full Face
Description: based on the subject's satisfaction questionnaire
Time Frame: Month 6
Population: only the 56 subjects who had provided answers in the subject's satisfaction questionnaire were included in the analysis
Measure: Number; unit: percentage of total subjects
Arm/Group | Azzalure and Restylane
Number analyzed (Participants) | 56
percentage of total subjects
  satisfied or very satisfied | 92.9
  neutral | 7.1

2. Secondary Outcome: Global Aesthetic Improvement From Baseline
Description: The scale responses are: -1 indicating "worse", 0 indicating "no change", 1 indicating "improved", 2 indicating "much improved" and 3 indicating "very much improved".
Time Frame: Week 3
Measure: Number; unit: percentage of total subjects
Arm/Group | Azzalure and Restylane
Number analyzed (Participants) | 60
percentage of total subjects
  Improved | 0
  Much or very much improved | 100

3. Secondary Outcome: Related Adverse Event
Description: Number of subjects reporting related adverse events
Time Frame: Month 6
Measure: Number; unit: participants
Arm/Group | Azzalure and Restylane
Number analyzed (Participants) | 60
participants | 14

ADVERSE EVENTS:
Arm/Group | Azzalure and Restylane
Serious Adverse Events (participants affected / at risk) | 2/60
Other Adverse Events (participants affected / at risk) | 18/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azzalure and Restylane (N=60)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral infarction (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azzalure and Restylane (N=60)
Injection site haematoma (General disorders) | 2 — administration site conditions
Nasopharyngitis (Infections and infestations) | 3
contusion (Injury, poisoning and procedural complications) | 2
headache (Nervous system disorders) | 2
Skin swelling (Skin and subcutaneous tissue disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less